CLINICAL TRIAL: NCT01488305
Title: Impact of Micronutrient Powders (MNP)With Homestead Food Production and an Intensive Community Level IYCF-BCC Intervention on Reducing Anemia and Improving Growth in Young Children, Nepal
Brief Title: Action Against Malnutrition Through Agriculture (AAMA) Plus MNP Study
Acronym: MNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 09-000076- AT; MNP impact study (Other Grant/Funding Number: 09-000076-AT10)
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2011-12

CONDITIONS: Anemia
Keywords: MNP; AAMA program; Nepal; HFP; IYCF; BCC
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Only government regular program (No Intervention): One arm is control arm, in this arm no additional program is added in government regular program
- AAMA arm (HFP and IYCF BCC) (Experimental): Second arm is AAMA project intervention which includes HFP activities, ENA and BCC activities
  Interventions: Other: AAMA project activities (HFP and IYCF BCC)
- MNP added in AAMA (Experimental): It is actually a intervention arm
  Interventions: Dietary Supplement: MNP (micro-nutrient powders); Other: AAMA project activities (HFP and IYCF BCC)

INTERVENTIONS:
Dietary Supplement: MNP (micro-nutrient powders) — MNP is added to explore the additional value of MNP in existing AAMA program
  Other Names: MNP sub study in AAMA
  Arms: MNP added in AAMA
Other: AAMA project activities (HFP and IYCF BCC) — This is the existing AAMA program
  Arms: AAMA arm (HFP and IYCF BCC); MNP added in AAMA

SUMMARY:
Helen Keller International (HKI), the ministry of health and population, and ministry of agriculture and cooperatives, of Nepal and local non-governmental organizations (NGO) partners are currently implementing a USAID funded Action Against Malnutrition Through Agriculture (AAMA) project in Baitadi district located in far Western development region of Nepal. HKI is undertaking this study within the AAMA project to test whether providing micro-nutrient powders (MNPs) in a programmatic context along with homestead food production (HFP) and an intensive community level Infant and Young Child Feeding Behavior change communication (IYCF-BCC) intervention will have a greater impact on reducing anemia and improving growth in young children than only providing the HFP and IYCF-BCC intervention without MNPs or a control with no intervention.

DETAILED DESCRIPTION:
The AAMA project uses the homestead food production (HFP) model that focuses on increasing households year round access to nutritious food as a platform to deliver a proven essential nutrition actions (ENA) related messages to household with children less than 2 years old. The AAMA project seeks to examine the effects of household level HFP on malnutrition. So the recipient and other partners wishes to undertake a study to explore a plausible delivery mechanism for MNPs along with HFP and intensive community level IYCF-BCC and their impact on infant/child growth and anemia.

The study is a cluster randomized controlled trial with a three arm factorial design. The trial involve 330 randomly selected children aged 6-9 months at the time of enrollment (n=110 per each of the three study arms). MNPs distributed through FCHVs to 110 children selected from communities that already have the HFP and IYCF-BCC intervention. This group of children will be compared on outcome parameters for anemia, growth (stunting, underweight and wasting) and infections (diarrhea, fever and cough) to a similar sub-set of children (n=110) who receive only the HFP and IYCF-BCC intervention and to a third sub-set of control children of similar age (n=110) who are not receiving either of these interventions. Children aged 6-9 months were chosen for the study because this age range captures the recommended age for introduction of complementary foods to children and our chosen age group also falls within the 0-24 month age range which is considered the period of rapid growth and development and therefore period of highest nutrient requirements in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-9 months of age during enrollment time
* Mothers who want to enroll their children in study

Exclusion Criteria:

* Severe anemia
* Children age below six months and age over 23 months during study time

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 334 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Anemia | One year
  All three arms anemia status will be compared after one year of MNP distribution (assess the additional value of MNP)

SECONDARY OUTCOMES:
Impact on growth of children | one year
  Assess the growth of children (wasting, underweigh and stunting)after one year of MNP distribution (MNP distribution started in March 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Pandey Rana, MPH, Principal Investigator — Helen Keller International
Locations (1):
- Helen Keller International, Nepal, Baitadī, Nepal

REFERENCES:
- See also: Helen Keller international — http://www.hki.org